CLINICAL TRIAL: NCT05253833
Title: A Phase 2, Randomized, Open-Label, Allopurinol-Controlled, Multicenter Study With Two Optional Extensions to Evaluate the Safety and Efficacy of AR882 Alone or in Combination With Allopurinol in Tophaceous Gout Patients
Brief Title: Phase 2 to Assess Efficacy and Safety in AR882 Alone or in Combination With Allopurinol in Patients With Tophaceous Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR882-203
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gout; Arthritis, Gouty; Hyperuricemia; Gout Chronic
MeSH Terms: conditions — Gout; Arthritis, Gouty; Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Allopurinol once daily for 24 weeks
  Interventions: Drug: Allopurinol Tablet
- Group 2 (Experimental): AR882 Dose 1 x 2 weeks, then Dose 2 x 22 weeks
  Interventions: Drug: AR882 Dose 1; Drug: AR882 Dose 2
- Group 3 (Experimental): AR882 Dose 1 + Allopurinol for 24 weeks
  Interventions: Drug: AR882 Dose 1; Drug: Allopurinol Tablet

INTERVENTIONS:
Drug: AR882 Dose 1 — Solid Oral Capsule
  Arms: Group 2; Group 3
Drug: AR882 Dose 2 — Solid Oral Capsule
  Arms: Group 2
Drug: Allopurinol Tablet — Solid tablet
  Arms: Group 1; Group 3

SUMMARY:
This study will assess the serum urate lowering effect, tophi reduction, and safety of AR882 alone and in combination with allopurinol in patients with tophaceous gout at two doses compared to allopurinol over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of gout
* at least 1 measurable tophus on the hands/wrists and/or feet/ankles ≥ 5 mm and ≤ 30 mm in the longest diameter.
* Patients who are NOT on approved ULT must have sUA > 7 mg/dL
* Patients who are on medically appropriate ULT must have sUA > 6 mg/dL
* Estimated Glomerular Filtration Rate (eGFR) ≥ 45 mL/min/1.73m2

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* Pregnant or breastfeeding
* History of kidney stones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 5 mg/dL at month 3 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 5 mg/dL at month 3

SECONDARY OUTCOMES:
Change from baseline in tophus area at Months 3 and 6 | 12 weeks and 24 weeks
  Comparison of the treatment groups for tophus area as measured by digital calipers
Change from baseline in tophus crystal volume at Months 6 | 24 weeks
  Comparison of the treatment groups for tophus crystal as measured by Dual-energy computerized tomography.
Serum urate (uric acid) (sUA) level <6, <4 and <3 mg/dL at month 3 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level <6, <4 and <3 mg/dL at month 3
Serum urate (uric acid) (sUA) level <6, < 5, <4 and <3 mg/dL at month 6 | 24 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level <6, < 5, <4 and <3 mg/dL at month 6
Incidence of Adverse Events | 24 weeks
  Treatment Emergent Adverse Events and Serious Adverse Event incidence.

CONTACTS AND LOCATIONS:
Overall Officials: R Keenan, MD, Study Chair — Arthrosi Therapeutics
Locations (12):
- United States (10):
  - Arthrosi Investigative Site (410), Birmingham, Alabama
  - Arthrosi Investigative Site (403), Phoenix, Arizona
  - Arthrosi Investigative Site (416), Sun City, Arizona
  - Arthrosi Investigative Site (417), Tucson, Arizona
  - Arthrosi Investigative Site (402), Tampa, Florida
  - Arthrosi Investigative Site (404), Boise, Idaho
  - Arthrosi Investigative Site (409), Ann Arbor, Michigan
  - Arthrosi Investigative Site (406), Greensboro, North Carolina
  - Arthrosi Investigative Site (408), Myrtle Beach, South Carolina
  - Arthrosi Investigative Site (401), Dallas, Texas
- Arthrosi Investigative Site (201), Auckland, New Zealand
- Arthrosi Investigative Site (303), Taichung, Taiwan